CLINICAL TRIAL: NCT04345627
Title: Japanese Lead Extraction Registry
Acronym: J-LEX
Status: Recruiting | Type: Observational
Sponsor: National Cerebral and Cardiovascular Center, Japan (Other)
Responsible Party: Principal Investigator, Kengo Kusano, Director of Cardiovascular Medicine, National Cerebral and Cardiovascular Center, National Cerebral and Cardiovascular Center, Japan
Other Study IDs: M29-146; UMIN000036078 (Other: UMIN-CTR)
Record Dates: First submitted 2020-04-10; First posted 2020-04-14 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Arrhythmia, Cardiac
Keywords: Lead extraction; Pacemaker; Defibrillator; Complication; REDCap
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Japanese Lead Extraction (J-LEX) Registry is an observational nationwide registry, performed by Japanese Heart Rhythm Society, collaborated with the National Cerebral and Cardiovascular Center. The acute success rate at discharge and the complications associated with transvenous lead extraction will be collected. J-LEX registry will provide a reliable information on indications, methods, the success rate, complications and the prognosis at 30 days prognosis.

DETAILED DESCRIPTION:
Japanese Lead Extraction (J-LEX) Registry is a nationwide, multicenter, observational registry, performed by Japanese Heart Rhythm Society, collaborated with National Cerebral and Cardiovascular Center. This study is a voluntary nationwide registry and data are collected prospectively using a Research Electronic Data Capture (REDCap) system until 30 days after the lead extraction. The investigators will collect the data regarding patient's background and lead characteristic, medical history, details about lead extraction procedure, lead characteristics, and outcomes. The data were anonymized in a linkable manner at each study site before they were sent. Based on the provided information, the annual incidence and predictive factors for outcome will be investigated by the event assessment committee.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing transvenous lead extraction in Japan.

Exclusion Criteria:

* Patients who receive open-chest surgical extraction alone.
* Patients who refused to consent.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Inpatients
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2018-07-01 (Actual); Primary Completion 2032-03-31 (Estimated); Study Completion 2032-03-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of procedural success | Through discharge from hospital, approximately up to 2 weeks.
  Procedural success was defined as complete or partial and is identified for each lead extracted.

SECONDARY OUTCOMES:
Number of in-hospital deaths | Through discharge from hospital, approximately up to 2 weeks.
  All-cause death, cardiovascular death, and procedure-related death
Number of patients with procedure-related complications | 4 weeks
  Bleeding events, embolic events, other all complications. Major bleeding events are defined according to Bleeding Academic Research Consortium criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Kengo Kusano, MD, PhD, Principal Investigator — National Cerebral and Cardiovascular Center, Japan
Locations (1):
- National Cerebral and Cardiovascular Center, Suita, Osaka, Japan